CLINICAL TRIAL: NCT01175408
Title: Blood Monitoring and Data Acquisition and Utilization in Patients With Type 2 Diabetes Treated With Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, Dr. Hugh Tildesley, Clinical Professor, Endocrine Research Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Monitoring and Acquisition T2D
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Remote Blood Glucose Monitoring System,; Continuous Glucose Monitoring System,; Self Monitoring Blood Glucose,; Strip Counting,; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Internet Intervention (Active Comparator): The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Interventions: Other: Remote Blood Glucose Monitoring
- Continuous Glucose Monitoring (Active Comparator): The use of CGMS (Sensor, receiver, transmitter) plus the uploading of results to the Internet-based software utility of CareLink Personal and generating reports that can be viewed and used at the patient's own preference. This group will send the data to their endocrinologist and receive feedback based on the uploaded glucose data.
  Interventions: Other: Continuous Glucose Monitoring
- SMBG (Active Comparator): The SMBG patients will be told that we are testing a new meter to check the accuracy of the meter. They will be asked to test at least 3 times a day and to keep a written diary of their sugar levels. The SMBG group will not know that we are counting strips and can not know about the SMBG With Knowledge group as it may bias the frequency that they test.
  Interventions: Other: SMBG
- SMBG With Knowledge (Active Comparator): The SMBG With Knowledge patients will be given a new meter and will be asked to test at least 3 times a day and to keep a written diary of their sugar levels. We will inform this group that we are measuring the frequency of SMBG testing.
  Interventions: Other: SMBG With Knowledge

INTERVENTIONS:
Other: Remote Blood Glucose Monitoring — The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Other Names: Internet Blood Glucose Monitoring System
  Arms: Internet Intervention
Other: Continuous Glucose Monitoring — The use of CGMS (Sensor, receiver, transmitter) (Medtronic Diabetes) plus the uploading of results to the Internet-based software utility of CareLink Personal and generating reports that can be viewed and used at the patient's own preference. This group will not receive feedback or suggestion based on the uploaded glucose data.
  Other Names: Sensors, CGMS
  Arms: Continuous Glucose Monitoring
Other: SMBG — The SMBG patients will be told that we are testing a new meter to check the accuracy of the meter. They will be asked to test at least 3 times a day and to keep a written diary of their sugar levels. The SMBG group will not know that we are counting strips and can not know about the SMBG With Knowledge group as it may bias the frequency that they test.
  Arms: SMBG
Other: SMBG With Knowledge — The SMBG With Knowledge patients will be given a new meter and will be asked to test at least 3 times a day and to keep a written diary of their sugar levels. We will inform this group that we are measuring the frequency of SMBG testing.
  Arms: SMBG With Knowledge

SUMMARY:
Management of type 2 diabetes is an ongoing challenge for patients and their doctors. In order to prevent complications, patients need to monitor and control their blood sugar levels. In addition, they may need to have an ongoing communication with their doctor in order to modify treatment. In this study the investigators wish to compare the benefits of continuous glucose monitoring system (CGMS) to an internet-based glucose monitoring system (IBGMS). The investigators also want to determine whether the frequency of blood glucose testing affects blood glucose control and to see whether the benefits of CGMS and IBGMS are independent of testing frequency.

DETAILED DESCRIPTION:
In this current study, the investigators wish to test several hypotheses: whether the frequency of SMBG is correlated with HbA1c, whether the knowledge that strips are being counted affects HbA1c, whether the reduction of HbA1c when using an IBGMS is independent of the frequency of testing, and whether there is a difference between IBGMS and CGMS in HbA1c reduction.

The investigators will recruit 100 patients with type 2 diabetes who satisfy the inclusion/exclusion criteria. For the first visit, the patients will be immediately randomized into four groups. One group will be testing 3 times a day (SMBG). The second group will be similar to the SMBG group except they will know that we are counting the frequency of testing (SMBG With Knowledge). The third group will use an IBGMS and the fourth group will use a CGMS. During the first visit, we will teach the patient how to use the programs and machinery for their group. All four groups will be asked to follow the protocol and to visit their doctor in 3 month intervals for 6 months along with completed laboratory blood test results.

For the SMBG and the SMBG With Knowledge group, each will be given a new meter and be asked to test 3 times a day. They will also be required to keep a diary of their SMBG levels. The difference between the two is that the SMBG With Knowledge group will know that we are counting strips. The SMBG group will believe that we are testing a new meter and will not know that the SMBG With Knowledge group exists. This deception is necessary to test the experimental effect of if the patient knows that we are counting the frequency of testing, does that affect the frequency that they are testing. The investigators will tell the SMBG group that we are testing the accuracy of a new meter and they should test 3 times a day.

For the CGMS and IBGMS group, they will also be counting the frequency of blood glucose testing to see whether the benefits from both are independent of the number of tests. Furthermore, we wish to compare the these two methods of blood glucose monitoring. Both groups will have to upload their data onto the internet and communicate with their doctor every 2 weeks using a secure online web site.

At the end of 3 and 6 months, we will collect the frequency of testing from each group to determine whether increased glycemic control correlates with increased testing. We will also collect their SMBG diaries to see whether the written data correlates with the data on their meter. The investigators will also be comparing a measure of their blood glucose levels for each group and determining the effectiveness of CGMS and IBGMS.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients being treated with insulin for at least 3 months HbA1c > 7%
* 25 years of age
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be trained on using the Continuous Glucose Monitoring System
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet Access on a Windows Personal Computer
* No prior use or training on CGMS in the past 6 months
* No prior use or training on IBGMS in the past 6 months

Exclusion Criteria:

Patients who do not meet the above criteria or are not willing to participate will not be included in the study. Additional exclusion criteria include:

* Patient with medical conditions that may affect their study participation or - - results will be excluded.
* Patients with the potential to become pregnant
* Patients using medications known to influence control of diabetes (eg steroids systemic or inhaled)
* Liver disease (AST or ALT levels > 2.5 times the reference level)
* Renal insufficient with a serum creatinine level > 200 μmol/L

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the A1c level or the change in A1c level | 6 Months

SECONDARY OUTCOMES:
A secondary endpoint includes adverse events such as unplanned hospitalizations for any cause that last more than 24 hours | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh D Tildesley, MD, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Klonoff DC, Bergenstal R, Blonde L, Boren SA, Church TS, Gaffaney J, Jovanovic L, Kendall DM, Kollman C, Kovatchev BP, Leippert C, Owens DR, Polonsky WH, Reach G, Renard E, Riddell MC, Rubin RR, Schnell O, Siminiero LM, Vigersky RA, Wilson DM, Wollitzer AO. Consensus report of the coalition for clinical research-self-monitoring of blood glucose. J Diabetes Sci Technol. 2008 Nov;2(6):1030-53. doi: 10.1177/193229680800200612. PMID 19885292
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] Yoo HJ, An HG, Park SY, Ryu OH, Kim HY, Seo JA, Hong EG, Shin DH, Kim YH, Kim SG, Choi KM, Park IB, Yu JM, Baik SH. Use of a real time continuous glucose monitoring system as a motivational device for poorly controlled type 2 diabetes. Diabetes Res Clin Pract. 2008 Oct;82(1):73-9. doi: 10.1016/j.diabres.2008.06.015. Epub 2008 Aug 12. PMID 18701183
- [Background] Tildesley HD, Mazanderani AB, Ross SA. Effect of Internet therapeutic intervention on A1C levels in patients with type 2 diabetes treated with insulin. Diabetes Care. 2010 Aug;33(8):1738-40. doi: 10.2337/dc09-2256. PMID 20668152